CLINICAL TRIAL: NCT06252948
Title: Gut Microbiome Studies in Patients With POEMS Syndrome and Other Plasma Cell Disorders
Acronym: Microbiome
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-013316; NCI-2022-10547 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Plasma Cell Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool donation will be requested from participants to assess gut microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- MULTIPLE MYELOMA at diagnosis GROUP: Multiple myeloma (before starting chemotherapy, radiation or stem cell transplant
  Interventions: Other: Non-interventional study (observational)
- Amyloid at diagnosis GROUP: AL amyloidosis (before starting chemotherapy or stem cell transplant)
  Interventions: Other: Non-interventional study (observational)
- Poems at diagnosis GROUP: POEMS at diagnosis (before starting chemotherapy, radiation, or stem cell transplant
  Interventions: Other: Non-interventional study (observational)
- Poems in Remission GROUP: POEMS in remission (no chemotherapy, radiation, or stem cell transplant for 2 years
  Interventions: Other: Non-interventional study (observational)
- MGUS GROUP: MGUS -not treated newly diagnosed
  Interventions: Other: Non-interventional study (observational)
- Health controls in same household GROUP: household member to be a healthy control (no chemotherapy or gastrointestinal illness to participate)
  Interventions: Other: Non-interventional study (observational)

INTERVENTIONS:
Other: Non-interventional study (observational) — Participants undergo stool sample collection, complete surveys, and have their medical record reviewed on study.
  Other Names: GMB

SUMMARY:
A Study to Evaluate Gut Microbiome with POEMS Syndrome and Other Plasma Cell Disorders

DETAILED DESCRIPTION:
The characteristics and role of gut microbiome rare plasma cell disorders- POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes) and amyloid light-chain (AL) amyloidosis, have not been explored; and their pathophysiology is quite elusive. To help understand rare plasma cell disorders and its association with gut microbiome, the investigators will study the stool samples of newly diagnosed POEMS patients and AL amyloidosis and compare it with patients with newly diagnosed monoclonal gammopathy of undetermined significance and multiple myeloma as well as healthy controls. Moreover, gut microbiome in newly diagnosed POEMS patients will be compared to POEMS patients in remission. It is the overall hypothesis that in POEMS patients the gut microbiome signature will differ between active disease (at diagnosis) and inactive disease (in remission), and the gut microbiome in POEMS patients will be different from patients with other plasma cell disorders and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with POEMS syndrome (newly diagnosed or in remission) or with newly diagnosed multiple myeloma (MM), monoclonal gammopathy of undetermined significance (MGUS), amyloid light chain (AL) amyloidosis or healthy controls from their households

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Substance abuse
* Antibiotics use or gastrointestinal endoscopy in the 3 months prior to the study participation
* Chronic gastrointestinal disorder
* Gastrointestinal surgeries in the past 2 years
* Chemotherapy (including anti-plasma cell treatment and steroids) or radiation treatment for cancer within the last 2 years or active cancer (other than plasma cell disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: POEMS Syndrome and Other Plasma Cell Disorders
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome characteristics in patients with POEMS syndrome and other plasma cell disorders | Baseline
  Stool samples will be collected by the patient using a stool self- collection kit provided to the participant by the study staff. Samples will be evaluated for characteristics of gut microbiome (α-diversity and β-diversity).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Gut microbiome (GMB) in patients with active POEMS syndrome will differ from POEMS patients with inactive disease. It will be also different from patients with other plasma cell disorders (amyloid light chain [AL] amyloidosis, multiple myeloma [MM] and monoclonal gammopathy of undetermined significance [MGUS]) and healthy controls.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials